CLINICAL TRIAL: NCT04151732
Title: Factors Associated With Future Fractures in Middle-aged Men and Women. A Prospective Cohort Study From Malmö Dietary Cancer Cohort
Brief Title: Factors Associated With Future Fractures in Middle-aged Men and Women
Acronym: MDCFract
Status: Completed | Type: Observational
Sponsor: Lund University (Other)
Collaborators: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: MDCFract1
Record Dates: First submitted 2019-10-24; First posted 2019-11-05 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Fractures, Bone; Fragility; Life Style
MeSH Terms: conditions — Fractures, Bone | interventions — Exercise; Ethanol; Tobacco Products; Heart Disease Risk Factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Physical activity, alcohol, tobacco — Physical activity, alcohol, tobacco - selfreported in the 1990's
Other: Hormonal factors — Hormonal factors - selfreported in the 1990's
Other: Cardiovascular disease — Cardiovascular disease - selfreported in the 1990's
Other: Anthropometric measures — Height, length, BMI

SUMMARY:
From prospectively collected health and life-style data and anthropometric data in the Malmo Diet and Cancer (MDC) cohort identify factors that predicts or are associated with forthcoming fracture in middle-aged men and women.

DETAILED DESCRIPTION:
In adults, the incidence of fractures increases with age. In predisposed individuals, even a minor trauma can result in a fracture. Such an injury is known as low-energy fracture or fragility fracture, and the risk increases with age. Fragility fractures may be preventable, either by changes in lifestyle or by medication of underlying diseases. Fragility fractures also put a burden both on the affected individual and on society. As the population age, more individuals are at risk, and the absolute numbers of fragility fractures increase. Therefore, identification of individuals at risk before fracture occurs would be ideal.In the prospectively collected Malmo Diet and Cancer (MDC) cohort a large number of health and life style variables have been gathered from randomly invited men and women in a city of 350,000 inhabitants in the 1990s'. The MDC database the investigators use for this study comprises 30,351 participants. Outcome is updated via crosslinking with the National Patient Register in Sweden.

MDC PhysFract - investigation of the following factors Socioeconomical factors: Level of education, employment status in middle age, physical activity / work load, living alone, stress, number of friends, feeling of loneliness.

Life style factors: Tobacco use, alcohol use. Summary of physical and psychological well-being.

MDC CardFract - investigation of the following factors Comorbidities: Hypertension, syncope/orthostatism, diabetes, coronary artery disease, atrial fibrillation, heart failure, ischemic stroke and others.

Pharmaceutical drugs associated with fracture risk. Cardiovascular blood tests.

MDC HormFract - investigation of the following factors Body composition: Weight at 20 yrs, weight change pattern, weight difference middle age minus 20 yrs.

Hormonal/gynecological status - women: Date for menarche and menopause, number of children, intake of oral contraceptives / hormonal replacement therapy, surgical menopause.

ELIGIBILITY:
Inclusion Criteria:

* Invited population based cohort from 1990's

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 30,351
Sampling Method: Non-Probability Sample
Enrollment: 30351 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Any fracture | 1992 - 2017
  Number of patients who suffered any fracture during follow-up (ICD-10 codes S12.x, S22.x, S32.x, S42.x, S52.x, S62.x, S32.x, S72.x, M48.4, M84.3, and M96.6)

SECONDARY OUTCOMES:
Multiple fractures | 1992 - 2017
  Number of patients who suffered multiple fractures during follow-up (ICD-10 codes S12.x, S22.x, S32.x, S42.x, S52.x, S62.x, S32.x, S72.x, M48.4, M84.3, and M96.6)
Death | 1992 - 2017
  Number of patients who died during follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Lund University / Skane university hospital, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moberg L, Hamrefors V, Fedorowski A, Rogmark C. Early menopause and weight loss are significant factors associated with risk of future fracture in middle-aged women. BMC Musculoskelet Disord. 2022 Aug 16;23(1):779. doi: 10.1186/s12891-022-05744-5. PMID 35974320
- [Derived] Rogmark C, Fedorowski A, Hamrefors V. Physical Activity and Psychosocial Factors Associated With Risk of Future Fractures in Middle-Aged Men and Women. J Bone Miner Res. 2021 May;36(5):852-860. doi: 10.1002/jbmr.4249. Epub 2021 Feb 18. PMID 33598954